CLINICAL TRIAL: NCT06258486
Title: Ultrasound Guided Inguinal Indocyanine Green Injection to Identify and Pre-emptively Seal Lymphatic Leaks
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICG lymphatic
Record Dates: First submitted 2024-01-24; First posted 2024-02-14 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Lymphocele; Prostate Cancer
MeSH Terms: conditions — Lymphocele; Prostatic Neoplasms | interventions — Prostatectomy

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into ICG versus no ICG injection after pelvic lymphadenectomy is completed.
Who Masked: Participant, Investigator
Masking Description: The investigator and participant will not know which arm the patient is randomized into while undergoing the surgery. It isn't until the surgery is complete that the patient will be randomized into either ICG injection versus not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ICG Injection (Experimental): This patient will undergo ICG injection into the lymph nodes in order to see if there are any leaks.
  Interventions: Drug: ICG injection; Procedure: Prostatectomy with pelvic lymph node dissection
- ICG non-injection (Placebo Comparator): This patient will not have ICG injection. the lymphadenectomy is considered complete at this point.
  Interventions: Other: Non-Injection/Control; Procedure: Prostatectomy with pelvic lymph node dissection

INTERVENTIONS:
Drug: ICG injection — Patient will have a green dye (ICG) injected into the lymph node to better visualize non-sealed leaks in order to pre-emptively seal any lymphatic leaks.
  Arms: ICG Injection
Other: Non-Injection/Control — No ICG injection
  Arms: ICG non-injection
Procedure: Prostatectomy with pelvic lymph node dissection — Robotic assisted prostatectomy with pelvic lymph node dissection

SUMMARY:
Goal is to determine whether intraoperative ICG injection can be used to identify and reduce formation of symptomatic lymphoceles in patients receiving robot-assisted prostatectomy.

DETAILED DESCRIPTION:
The goal of this clinical trial is to determine whether intraoperative ICG injection can be used to identify and reduce formation of symptomatic lymphoceles in patients receiving robot-assisted prostatectomy. The main question is if it could improve patients' quality of life and infection risk post-surgery. It would also help to decrease emergency room visits as well as additional procedures. Researchers will compare those who receive the ICG and those who do not.

Patients will be randomized into the ICG arm versus no ICG arm after pelvic lymphadenectomy is done.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing robotic assisted laparoscopic lymph node dissection

Exclusion Criteria:

* Patient not undergoing extended lymph node dissection
* History of allergy to iodides

Ages: 45 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Drain output <100 mL | 2 weeks
  A sample of 12 recent patients receiving the current standard procedure had a mean drain volume for the first 24 hours of 218 mL and standard deviation of 102. With a hoped-for reduction to <100 mL/ 24 hr mean in the treatment arm, there would be 99% power to detect a difference, and 80% power to detect a difference of 57 mL between treatment and control arms. Given the small sample used for this power estimate, we believe that it is appropriate to power for a range of potential standard deviations and potential differences.

SECONDARY OUTCOMES:
Lymphocele formation | 4 weeks
  Any lymphocele formation will be logged; any lymphocele proven by imaging

CONTACTS AND LOCATIONS:
Overall Officials: David Finley, MD, Principal Investigator — Kaiser Permanente

IPD SHARING:
Plan to Share IPD: No
No indication to share individual participant data with other researchers.

REFERENCES:
- [Result] Motterle G, Morlacco A, Zanovello N, Ahmed ME, Zattoni F, Karnes RJ, Dal Moro F. Surgical Strategies for Lymphocele Prevention in Minimally Invasive Radical Prostatectomy and Lymph Node Dissection: A Systematic Review. J Endourol. 2020 Feb;34(2):113-120. doi: 10.1089/end.2019.0716. PMID 31797684
- [Result] Tewari A, Sooriakumaran P, Bloch DA, Seshadri-Kreaden U, Hebert AE, Wiklund P. Positive surgical margin and perioperative complication rates of primary surgical treatments for prostate cancer: a systematic review and meta-analysis comparing retropubic, laparoscopic, and robotic prostatectomy. Eur Urol. 2012 Jul;62(1):1-15. doi: 10.1016/j.eururo.2012.02.029. Epub 2012 Feb 24. PMID 22405509
- [Result] Tsaur I, Thomas C. Risk factors, complications and management of lymphocele formation after radical prostatectomy: A mini-review. Int J Urol. 2019 Jul;26(7):711-716. doi: 10.1111/iju.13964. Epub 2019 Apr 2. PMID 30939628
- [Result] Gloger S, Ubrig B, Boy A, Leyh-Bannurah SR, Siemer S, Arndt M, Stolzenburg JU, Franz T, Oelke M, Witt JH. Bilateral Peritoneal Flaps Reduce Incidence and Complications of Lymphoceles after Robotic Radical Prostatectomy with Pelvic Lymph Node Dissection-Results of the Prospective Randomized Multicenter Trial ProLy. J Urol. 2022 Aug;208(2):333-340. doi: 10.1097/JU.0000000000002693. Epub 2022 Apr 15. PMID 35422136